CLINICAL TRIAL: NCT04241926
Title: Single-lumen 5Fr and Triple-lumen 6Fr PICCs Are Accurate for Hemodynamic
Brief Title: Single-lumen 5Fr and Triple-lumen 6Fr PICCs Are Accurate for Hemodynamic Measurement by Transpulmonary Thermodilution.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Antonio Maria Dell Anna (Unknown); Sofia Cacciola (Unknown); Claudio Sandroni (Unknown); Giulia Chiuri (Unknown); Mauro Pittiruti (Unknown); Cesare Colosimo (Unknown); Maria Giuseppina Annetta (Unknown); Massimo Antonelli (Unknown)
Responsible Party: Principal Investigator, Dr.ssa Sonia D'Arrigo, Medical Doctor - PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PICC 5Fr and 6Fr-CICC for TPTD
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Peripherally Inserted Central Catheters; Centrally Inserted Central Catheter; Transpulmonary Thermodilution; Hemodynamic Monitoring
Keywords: PICC; CICC; Cardiac output; shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transpolmonary thermodilution — Thermodilution was attempted via PICC and via CICC in the same patient

SUMMARY:
Peripherally inserted central catheters (PICCs) are increasingly used in intensive care unit (ICU) as an alternative to centrally inserted central catheters (CICCs) for intravenous infusion. In the present study the investigators try to assess their reliability for measuring cardiac index (CI) with trans-pulmonary thermodilution (TPTD) technique.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years) admitted to the ICU
* Patients requiring hemodynamic monitoring using EV1000TM
* Patients having both PICC and CICC in place (these patients had their PICC replaced with a CICC, usually at the time of ICU admission, or vice versa, usually at the end of their ICU stay, and were enrolled immediately after the placement of the new device before the previous one was removed)

Exclusion Criteria:

* body weight <40 kg
* severe aortic regurgitation or intra-cardiac shunt
* treatment with an intra-aortic balloon pump
* contraindication for placement of PICC, CICC or a femoral arterial catheter
* abdominal aneurism
* extracorporeal circulation
* pregnancy
* lack of informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Cardiac Index comparison via PICC | one hour
  comparison of hemodynamic measurements made by the TPTD from the VolumeView/EV1000TM system via PICC vs. CICC.

SECONDARY OUTCOMES:
Comparison of single-lumen 5Fr PICCs to CICC | one hour
  Comparison of single-lumen 5 Fr PICCs to CICC in their reliability of assessing cardiac output
Comparison of triple-lumen 6Fr PICCs to CICC | one hour
  Comparison of triple-lumen 6 Fr PICCs to CICC in their reliability of assessing cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Study Chair — Università Cattolica del sacro Cuore- Fondazione Policlinico Universitario A. Gemelli IRCSS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Arrigo S, Sandroni C, Cacciola S, Dell'Anna AM, Pittiruti M, Annetta MG, Colosimo C, Antonelli M. Are single-lumen 5Fr and triple-lumen 6Fr PICCs suitable for hemodynamic assessment by trans-pulmonary thermodilution? A pilot study. Ann Intensive Care. 2020 Dec 7;10(1):165. doi: 10.1186/s13613-020-00785-2. PMID 33284392